CLINICAL TRIAL: NCT06654635
Title: Comparison Between Ultrasound Guided Rhomboid Intercostal Plane Block and Thoracic Erector Spinae Plane Block in Patients Undergoing Upper Abdominal Surgery: A Randomized Controlled Trial
Brief Title: Ultrasound Guided Rhomboid Intercostal Plane Block Versus Thoracic Erector Spinae Plane Block in Upper Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Omima Mohammed Fakher Eldin Ali, Assistant Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264MD87/5/23
Record Dates: First submitted 2024-10-22; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Ultrasound; Rhomboid Intercostal Plane Block; Thoracic Erector Spinae Plane Block; Upper Abdominal Surgery
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Rhomboid intercostal plane block group (Experimental): The patients in this group will receive ultrasound -guided rhomboid intercostal plane block after induction of general anesthesia. The rhomboid intercostal block will be performed at the T6 levels, bilaterally.
  Interventions: Drug: Rhomboid intercostal plane block
- Erector spinae plane block group (Experimental): The patients in this group will receive ultrasound -guided Erector spinae plane block after induction of general anesthesia. ESP block will be performed at the level of T9 bilaterally.
  Interventions: Other: Erector spinae plane block
- Control group (Experimental): No block will be performed, and patient will receive general anesthesia (GA) only.
  Interventions: Other: Control group

INTERVENTIONS:
Drug: Rhomboid intercostal plane block — The patients in this group will receive ultrasound -guided rhomboid intercostal plane block after induction of general anesthesia. The rhomboid intercostal block will be performed at the T6 levels, bilaterally.
  Arms: Rhomboid intercostal plane block group
Other: Erector spinae plane block — The patients in this group will receive ultrasound -guided Erector spinae plane block after induction of general anesthesia. Erector spinae plane block will be performed at the level of T9 bilaterally.
  Arms: Erector spinae plane block group
Other: Control group — No block will be performed, and patient will receive general anesthesia (GA) only.
  Arms: Control group

SUMMARY:
The aim of the work is to evaluate the analgesic efficacy of ultrasound guided rhomboid intercostal plane block versus ultrasound guided thoracic erector spinae block in patients undergoing upper abdominal surgery.

DETAILED DESCRIPTION:
Abdominal surgery is one of the most definitive and mainstay treatment options for abdominal pathologies in clinical practice. Acute postoperative pain is a major challenge in the postoperative period.

The improved safety and efficacy that ultrasound brings to regional anesthesia helped promote its use and realize the benefits that regional anesthesia has over general anesthesia, such as decreased morbidity and mortality, superior postoperative analgesia, cost-effectiveness, decrease postoperative complications and an improved postoperative course .

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 21-65 years.
* Both gender.
* American Society of Anesthesiologists (ASA) classification I-II.
* Presented for elective upper abdominal surgery.

Exclusion Criteria:

* Patients refused to participate.
* Patients with known or suspected allergy to the used medication.
* Patients with preoperative chronic pain.
* Patients with major cardiac, renal, respiratory, or hepatic disease.
* Patients with potential risk of coagulopathy.
* Obese patients with body mass index (BMI) >35.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia will be provided in the form of IV morphine 3 mg boluses if the patient indicates The visual analogue scale (VAS). ≥ 4 with maximum dose 20 mg for 24 hours. The total amount of morphine (mg) given will be recorded for the 3 groups.

SECONDARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  Postoperative pain will be assessed by visual analogue scale (VAS) 30 min from admission to PACU, 2, 4, 6, 12, 18 and 24 h postoperative (0= no pain, 10= sever pain).
Time to 1st request of rescue analgesia | 24 hours postoperatively
  Time to 1st request for the rescue of analgesia (time from the end of surgery till first dose of morphine administrated ) will be recorded.
Heart rate | Every 15 min till the end of surgery
  Heart rate will be measured preoperative, after induction, after receiving block and every 15 min till the end of surgery
Mean arterial blood pressure | Every 15 min till the end of surgery
  Mean arterial blood pressure will be measured preoperative, after induction, after receiving block and every 15 min till the end of surgery
Incidence of side effects | 24 hours Postoperatively
  Any undesirable adverse events will be treated and recorded (e.g., bradycardia, hypotension, pneumothorax, hematoma, nerve injury and nausea, vomiting, local anesthetic systemic toxicity (LAST), respiratory depression or any other complication).

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.